CLINICAL TRIAL: NCT03526237
Title: Novel Intervention Linking Public Housing With Primary Care to Prevent Diabetes
Acronym: SHAPE-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 00036688; 1R34DK097724 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-05-16 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus Risk; Obesity; Cardiovascular Risk Factor
Keywords: diabetes; prevention; risk; obesity; weight loss; community based
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The 24-week treatment (Experimental): The 24-week treatment, Sisters Health And Primary CarE Uniting and Preventing Diabetes (SHAPE UP) 12 weekly peer group (adapted Group Lifestyle Balance Program) sessions followed by 3 monthly group maintenance sessions held in Public Housing locations; b) Individual coaching and patient activation during 24 week period; 2) Community Outreach Care Coordination: Referral, navigation assistance, patient activation, and cross-linkage to FQHC services.
  Interventions: Behavioral: 24 week community based DPP Group Lifestyle Balance Program
- Wait-list Control (Other): Control arm participants will receive: 1) Usual care in FQHC/primary care clinic 2) Individual counseling about pre-diabetes risk at baseline; mailed written NIDDK patient education materials (weight loss, physical activity, nutrition) at weeks 6, 12, 18; 2) At the end of the 24 week intervention, the wait list control arm will be invited to participate and receive the group based DPP sessions.
  Interventions: Behavioral: Wait-List Control community based DPP Group Lifestyle Balance Program

INTERVENTIONS:
Behavioral: 24 week community based DPP Group Lifestyle Balance Program — a) 12 weekly peer group (adapted Group Lifestyle Balance Program) sessions followed by 3 monthly group maintenance sessions held in Public Housing locations; b) Individual coaching and patient activation during 24 week period; 2) Community Outreach Care Coordination: Referral, navigation assistance, patient activation, and cross-linkage to FQHC services.
  Arms: The 24-week treatment
Behavioral: Wait-List Control community based DPP Group Lifestyle Balance Program — Control arm participants will receive: 1) Usual care in FQHC/primary care clinic 2) Individual counseling about pre-diabetes risk at baseline; mailed written NIDDK patient education materials (weight loss, physical activity, nutrition) at weeks 6, 12, 18; 2) At the end of the 24 week intervention, the wait list control arm will be invited to participate and receive the group based DPP sessions.
  Arms: Wait-list Control

SUMMARY:
(Sisters Health And Primary CarE Uniting and Preventing Diabetes; aka SHAPE UP) will consist of: 1) Neighborhood DPP Intervention: group DPP sessions and individual coaching; 2) Preventive Care Coordination to FQHC: referral, navigation assistance, patient activation, linkage to primary care (community initiated referrals) and linkage to DPP program (FQHC initiated referrals)

DETAILED DESCRIPTION:
SHAPE-UP we will use a randomized between groups wait-list design wherein the experimental treatment will be compared to best practices FHCN/FQHC services waitlist control (with an educational supplement for control). At the 24-week point, the waitlist control participants will be invited to receive the intervention. This combines a between groups RCT design with a phase change/within-group design for maximum efficiency with a limited N. Randomization will occur at the level of the individual participant. To sustain participant interest and to address obesity-related needs, control arm participants will receive Best Practices services including 1) Individual counseling about pre-diabetes risk at baseline; 2) mailed written materials at weeks 6, 12, 18; and 3) As needed additional FQHC Primary Care services (as mentioned, referral to the DPP obesity intervention and FHCN/FQHC primary care services will be bidirectional. The RE-AIM framework will guide process and impact evaluation measures of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age or older
2. Body-mass index of > 25 kg/m2 or waist circumference >35 inches
3. ADA diabetes risk assessment > at risk for pre-diabetes
4. Casual capillary blood glucose > 110 mg/dl <200
5. Access to phone
6. Resident in or surrounding partnering Public Housing neighborhood and eligible for FHCN services

Exclusion Criteria:

1. Exclusions for diseases likely to limit lifespan and/or increase risk of interventions: a) Cancer requiring treatment in the past 5 years; b) Cardiovascular disease: "Yes" response to any item on the modified Physical Activity Readiness Questionnaire; Uncontrolled hypertension: SBP >180 mmHg or DBP >105 mmHg; Heart attack, stroke, or transient ischemic attack in the past 6 months; c) Lung disease: Chronic obstructive airways disease or asthma requiring home oxygen
2. Exclusions related to metabolism: a) Diabetes at baseline; b) Casual capillary blood glucose >200 mg/dl; c) History of anti-diabetic medication use (oral agents or insulin) except during gestational diabetes; d) Pregnant female; e) Self-report of disease associated with disordered glucose metabolism: Cushing's syndrome; acromegaly; pheochromocytoma; chronic pancreatitis
3. Exclusion for conditions or behaviors likely to affect the conduct of the study: a) Unable or unwilling to provide informed consent; b) Unable to read written English

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change in BMI | Wk. 12 and 24
  weight and height will be combined to report BMI in kg/m^2)

SECONDARY OUTCOMES:
Change in Waist circumference | Wk 12 and 24
  waist (abdominal) circumference in centimeters
Change in Lipids (LDL, HDL, Total Cholesterol and Triglycerides) | Wk. 12 and 24
  Measured using a capillary blood sample Cholestech LDX
Change in A1C | Wk 12 and 24
  Measured using a capillary blood sample DCA 2000 analyzer
Change in Diet and exercise Behaviors | Wk 12 and 24
  Assessed by the Health Promoting Lifestyle Profile II

CONTACTS AND LOCATIONS:
Overall Officials: Gayenell S Magwood, PhD, Principal Investigator — Medical University of South Carolina